CLINICAL TRIAL: NCT02288325
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Relapse-Prevention Study With Levomilnacipran ER in Patients With Major Depressive Disorder
Brief Title: A Multicenter, Relapse Prevention Study With Levomilnacipran Extended Release (ER) in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVM-MD-15
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-09

CONDITIONS: Depressive Disorder, Major
Keywords: Fetzima; Relapse-prevention; Placebo-controlled
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open-Label FETZIMA® (Experimental): FETZIMA® (levomilnacipran extended release [ER]) taken orally during flexible dose titration up to 40, 80 or 120 mg once daily in 8-week run-in period followed by fixed dose of 40, 80 or 120 mg once daily in 12-week stabilization period.
  Interventions: Drug: Levomilnacipran ER
- Double-Blind Placebo (Placebo Comparator): Dose-matched placebo taken orally once daily for 26 weeks during double-blind treatment period.
  Interventions: Drug: Placebo
- Double-Blind FETZIMA® (Experimental): FETZIMA® (levomilnacipran ER) taken orally at fixed dose of 40, 80 or 120 mg once daily for 26 weeks during double-blind treatment period.
  Interventions: Drug: Levomilnacipran ER

INTERVENTIONS:
Drug: Levomilnacipran ER — Levomilnacipran ER taken orally at 40, 80 or 120 mg once daily.
  Other Names: FETZIMA®
  Arms: Double-Blind FETZIMA®; Open-Label FETZIMA®
Drug: Placebo — Dose-matched placebo taken orally once daily.
  Arms: Double-Blind Placebo

SUMMARY:
This study evaluates the efficacy, safety and tolerability of levomilnacipran extended-release (ER) compared with placebo in the prevention of depression relapse in major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria

* Currently meet the DMS-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th edition) criteria for Major Depressive Disorder (MDD)
* The participant must have an ongoing major depressive episode of at least 8 weeks and no more than 18 months
* The participant must have at least 3 lifetime episodes of MDD (including the current episode)

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not practicing a reliable method of birth control
* Participants who are considered a suicide risk
* History of non-response to 2 or more antidepressants (after adequate treatment)
* Participants who have a history of meeting DMS-5 criteria for manic, hypomanic, or mixed episode, obsessive-compulsive disorder, schizophrenia or other psychotic disorder
* Panic disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Migliore, Study Director — Forest Research Institute, Inc., an affiliate of Allergan, plc
Locations (47):
- United States (47):
  - Forest Investigative Site 053, Birmingham, Alabama
  - Forest Investigative Site 050, Dothan, Alabama
  - Forest Investigative Site 039, Phoenix, Arizona
  - Forest Investigative Site 048, Beverly Hills, California
  - Forest Investigative Site 047, Chino, California
  - Forest Investigative Site 028, Costa Mesa, California
  - Forest Investigative Site 021, Encino, California
  - Forest Investigative Site 052, Lemon Grove, California
  - Forest Investigative Site 042, Oceanside, California
  - Forest Investigative Site 016, Sherman Oaks, California
  - Forest Investigative Site 037, Sherman Oaks, California
  - Forest Investigative Site 043, Simi Valley, California
  - Forest Investigative Site 040, Cromwell, Connecticut
  - Forest Investigative Site 038, Norwich, Connecticut
  - Forest Investigative Site 023, Bradenton, Florida
  - Forest Investigative Site 018, Fort Myers, Florida
  - Forest Investigative Site 001, Jacksonville, Florida
  - Forest Investigative Site 008, Jacksonville Beach, Florida
  - Forest Investigative Site 057, Kissimmee, Florida
  - Forest Investigative Site 009, Orlando, Florida
  - Forest Investigative Site 045, West Palm Beach, Florida
  - Forest Investigative Site 034, Alpharetta, Georgia
  - Forest Investigative Site 049, Smyrna, Georgia
  - Forest Investigative Site 019, Schaumburg, Illinois
  - Forest Investigative Site 020, Methuen, Massachusetts
  - Forest Investigative Site 051, Watertown, Massachusetts
  - Forest Investigative Site 044, Cherry Hill, New Jersey
  - Forest Investigative Site 031, Brooklyn, New York
  - Forest Investigative Site 036, Cedarhurst, New York
  - Forest Investigative Site 013, Mount Kisco, New York
  - Forest Investigative Site 003, New York, New York
  - Forest Investigative Site 005, New York, New York
  - Forest Investigative Site 055, Rochester, New York
  - Forest Investigative Site 058, Charlotte, North Carolina
  - Forest Investigative Site 011, Dayton, Ohio
  - Forest Investigative Site 035, Tulsa, Oklahoma
  - Forest Investigative Site 046, Portland, Oregon
  - Forest Investigative Site 041, Salem, Oregon
  - Forest Investigative Site 012, Media, Pennsylvania
  - Forest Investigative Site 030, Memphis, Tennessee
  - Forest Investigative Site 033, Memphis, Tennessee
  - Forest Investigative Site 054, Dallas, Texas
  - Forest Investigative Site 059, Houston, Texas
  - Forest Investigative Site 014, Murray, Utah
  - Forest Investigative Site 010, Charlottesville, Virginia
  - Forest Investigative Site 056, Roanoke, Virginia
  - Forest Investigative Site 026, Brown Deer, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Run-in Period
Arm/Group | Open-Label FETZIMA® | Double-Blind Placebo | Double-Blind FETZIMA®
Started | 644 | 0 | 0
Completed | 499 | 0 | 0
Not Completed | 145 | 0 | 0
Not completed — Adverse Event | 48 | 0 | 0
Not completed — Lack of Efficacy | 16 | 0 | 0
Not completed — Withdrawal of Consent | 28 | 0 | 0
Not completed — Lost to Follow-up | 25 | 0 | 0
Not completed — Protocol Violation | 17 | 0 | 0
Not completed — Non-Compliance With Study Drug | 3 | 0 | 0
Not completed — Reason not Specified | 8 | 0 | 0
Period: Stabilization Period
Arm/Group | Open-Label FETZIMA® | Double-Blind Placebo | Double-Blind FETZIMA®
Started | 429 (70 participants did not enter Stabilization Period (69 did not meet entry criteria; 1 other reason)) | 0 | 0
Completed | 331 | 0 | 0
Not Completed | 98 | 0 | 0
Not completed — Adverse Event | 13 | 0 | 0
Not completed — Lack of Efficacy | 22 | 0 | 0
Not completed — Withdrawal of Consent | 23 | 0 | 0
Not completed — Lost to Follow-up | 12 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 0
Not completed — Non-Compliance With Study Drug | 5 | 0 | 0
Not completed — Reason not Specified | 15 | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | Open-Label FETZIMA® | Double-Blind Placebo | Double-Blind FETZIMA®
Started | 0 | 159 (7 participants did not enter Double-Blind Period (2 did not meet entry criteria; 5 other reasons)) | 165 (7 participants did not enter Double-Blind Period (2 did not meet entry criteria; 5 other reasons))
Completed | 0 | 135 | 139
Not Completed | 0 | 24 | 26
Not completed — Adverse Event | 0 | 2 | 5
Not completed — Withdrawal of Consent | 0 | 8 | 8
Not completed — Lost to Follow-up | 0 | 4 | 5
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Non-Compliance With Study Drug | 0 | 1 | 4
Not completed — Multiple Reasons | 0 | 8 | 2

BASELINE CHARACTERISTICS:
Population: Run-in Phase (RIP) Safety Population comprised all participants in the screened population who took at least 1 dose of open-label levomilnacipran during the RIP.
Arm/Group | Open-Label FETZIMA®
Number analyzed (Participants) | 644
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 404
  Male | 240

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse During the Double-Blind Treatment Period (DBTP)
Description: Time to relapse for the median was measured in days from randomization date at the start of the DBTP to relapse date during DBTP. Relapse was defined as meeting any 1 or more of the following criteria: 1) Insufficient therapeutic response at any one visit, including a >/= 2 increase in Clinical Global Impressions-Severity (CGI-S) score (range 1 to 7) compared with that obtained at randomization, or risk of suicide as determined by the investigator, or need for hospitalization due to worsening of depression as determined by the investigator, or need for alternative treatment of depressive symptoms as determined by the Investigator; 2) Montgomery-Asberg Depression Rating Scale (MADRS) total score >/= 18 (range 0 to 60) at 2 consecutive visits (second visit within 7 to 14 days after the first visit at which the MADRS total score was ≥ 18). Participant was considered censored at the last visit during DBTP if participant did not meet the relapse criteria during DBTP.
Time Frame: From the randomization date (Week 20) to the relapse date during the 26-week DBTP (up to Week 46)
Population: Double-blind Intent-to-Treat (ITT) population comprised of all participants in the Double-blind Safety Population who had at least 1 post-randomization assessment of MADRS or those participants who met relapse criteria during the DBTP of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Double-Blind Placebo | Double-Blind FETZIMA®
Number analyzed (Participants) | 159 | 165
days | NA [NA to NA] — Not available due to insufficient number of events. | NA [NA to NA] — Not available due to insufficient number of events.
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind FETZIMA®; Test type: Superiority; p = 0.0212, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.33 to 0.92]

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Arm/Group | Open-Label FETZIMA® | Double-Blind Placebo | Double-Blind FETZIMA®
All-Cause Mortality (participants affected / at risk) | 0/644 | 0/159 | 0/165
Serious Adverse Events (participants affected / at risk) | 9/644 | 1/159 | 2/165
Other Adverse Events (participants affected / at risk) | 430/644 | 29/159 | 41/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label FETZIMA® (N=644) | Double-Blind Placebo (N=159) | Double-Blind FETZIMA® (N=165)
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label FETZIMA® (N=644) | Double-Blind Placebo (N=159) | Double-Blind FETZIMA® (N=165)
Nausea (Gastrointestinal disorders) | 174 | 5 | 13
Constipation (Gastrointestinal disorders) | 69 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 37 | 2 | 0
Headache (Nervous system disorders) | 103 | 12 | 17
Dizziness (Nervous system disorders) | 50 | 4 | 1
Heart rate increased (Investigations) | 71 | 4 | 4
Blood pressure increased (Investigations) | 36 | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 57 | 2 | 1
Tachycardia (Cardiac disorders) | 50 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 46 | 10 | 16
Insomnia (Psychiatric disorders) | 34 | 2 | 5
Nasopharyngitis (Infections and infestations) | 25 | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.